CLINICAL TRIAL: NCT02544555
Title: Safety and Efficacy of Subintimal Versus Intraluminal Approach for Atherosclerotic Chronic Occlusive Femoro-Popliteal Arterial Disease: Prospective, Multicenter, Randomized, Controlled Trial (SCENARIO-FP)
Brief Title: Efficacy of Subintimal vs Intraluminal Approach for Atherosclerotic Chronic Occlusive Femoropopliteal Arterial Disease
Acronym: SCENARIO-FP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seung Woon Rha, Clinical Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCENARIO-FP
Record Dates: First submitted 2015-08-27; First posted 2015-09-09 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Arterial Disease; Atherosclerosis
Keywords: Peripheral arterial disease; Atherosclerosis; Intraluminal approach; Subintimal approach
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intentional intraluminal approach (Experimental): Intentional intraluminal approach is the way that the passage of guidewire in chronic total occlusive femoro-popliteal arterial lesion is performed via intraluminal route using various intraluminal devices. in an intraluminal approach, the response to the balloon is more favorable, but the outcome depends on the experience of the surgeon, and the approach requires more time and is more costly.
  Interventions: Procedure: Intentional intraluminal approach
- Intentional subintimal approach (Active Comparator): Intentional subintimal approach is the method that recanalization is performed via subintimal route with a 0.035-inch looped guidewire and a supporting catheter at the occlusion site. Due to its simplicity and low cost, this approach has been used for many patients with femoropopliteal occlusion.
  Interventions: Procedure: Intentional subintimal approach

INTERVENTIONS:
Procedure: Intentional intraluminal approach — Interventionist performs intentional intraluminal approach to angioplasty. Dedicated 018 and 014 guidewire for Chronic Total Occlusion (CTO) lesion and Chronic Total Occlusion (CTO) devices such as Truepath or Frontrunner can be chosen by interventionist. Methods to confirm successful intraluminal wiring will be selected, as follows; 1) examination for guidewire position in different two angles on fluoroscopy or 2) intravascular ultrasound (IVUS) exam after predilation is performed with an appropriately sized angioplasty balloon. After the guidewire is passed through the lumen of target lesion, predilation of the target lesion with an optimally sized balloon will be performed prior to stent implantation. Provisional stenting should be performed, if the case that optimal ballooning response is not obtained.
  Arms: Intentional intraluminal approach
Procedure: Intentional subintimal approach — Interventionist performs Intentional subintimal approach to angioplasty. 035 Terumo guidewires will be used. If 035 Terumo guidewire is not able to re-entry, Re-entry devices such as Offroad or OUTBACK catheter can be used. After the guidewire is passed through the subintimal layer of target lesion, predilation of the target lesion with an optimally sized balloon will be performed prior to stent implantation. Provisional stenting should be performed; the case that optimal ballooning response is not obtained should be enrolled. The sub-optimal balloon response is defined as a residual pressure gradient of >15 mmHg, residual stenosis of >30%, and flow-limiting dissection.
  Arms: Intentional subintimal approach

SUMMARY:
There are two ways of approaching atherosclerotic chronic occlusive femoro-popliteal arterial lesion with guide wire. One is the intraluminal approach of passing guide wire through the atheroma, the other is the subintimal approach of passing wire through the subintima of the vessel.

Either of these two interventional technique can be chosen depending on the character of the lesions they have their own pros and cons which affects the success of the intervention. The study is limited to retrospective studies to which interventional technique is better for post-procedural recurrence rate, however there is no prospective randomized controlled study.

DETAILED DESCRIPTION:
During interventions for atherosclerotic femoro-popliteal arterial lesion, chronic occlusive lesions are commonly encountered. The decision to approach these lesions by either guide wire, intraluminal approach or subintimal approach is by the decision of the operator. The subintimal approach intentionally passes the guide wire through the subintimal layer of vessel which was developed by Dr. Bolia. Through the subintimal approach, the success rate of procedure has increased. However this technique has shown some limitations which are guide wire re-entry, intimal injury, lengthening of the original lesion, periadventitial hematoma, perforated vessel, collateral vascular occlusion and limited usage of atherectomy devices.

On the contrary, intimal approach is not only able to overcome the limitations of the subintimal approach, but it has shown an advantage in improving the success rate of the procedure by the variable techniques of anterograde, retrograde and trans-collaterals approach. These techniques however usually require longer procedure time with more exposure to larger amounts of intravenous contrast and radiation. It often cause the need for more interventional devices which results in higher expense such that it is a less cost-effective method.

Recently the recommendation is the combination of these 2 interventional techniques depending on the character of lesions. As above, these approaches are chosen depending on the character of the lesion, however there are only limited retrospective studies without prospective randomized controlled study present to decide which method is better in terms of post-procedural recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Criteria

  1. Age 20 years of older
  2. Symptomatic peripheral-artery disease with (Rutherford 2 - 6); moderate to severe claudication (Rutherford 2-3), chronic critical limb ischemia with pain while at rest (Rutherford 4), or with ischemic ulcers (Rutherford 5-6)
  3. Patients with signed informed consent
* Anatomical Criteria

  1. Chronic occlusive lesion in coronary angiography
  2. Stenosis of <50% atherosclerotic lesion of the ipsilateral femoropopliteal artery
  3. Residual stenosis of <50% atherosclerotic lesion of the ipsilateral femoro-popliteal artery after treatment for >50% of the lesion.
  4. Patent (≤50% stenosis) ipsilateral iliac artery or concomitantly treatable ipsilateral iliac lesions (≤30% residual stenosis), At least one patent (less than 50% stenosed) tibioperoneal run-off vessel.
  5. Only balloon angioplasty can be performed for popliteal arterial lesion, however if suboptimal or bailout result is expected with sole balloon angioplasty, stent placement is allowed. Bailout or suboptimal result is defined as SFA lesion.

Exclusion Criteria:

1. Under 20 years-old or over 85 years-old.
2. Disagree with written informed consent
3. Major bleeding history within prior 2 months
4. Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, cilostazol, or contrast agent
5. Acute limb ischemia
6. Previous bypass surgery or stenting of the ipsilateral femoro-popliteal artery
7. Untreated inflow disease of the ipsilateral pelvic arteries (more than 50% stenosis or occlusion)
8. Patients with major amputation ("above the ankle" amputation) which has been done, is planned or required
9. Patients with life expectancy <1 year due to comorbidity
10. Severe medical or surgical illness limit participating study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
The rate of binary restenosis. | One year
  the rate of binary restenosis (stenosis of at least 50 percent of the luminal diameter) or PSVR ≥ 2.5 or zero (PSVR=peak systolic velocity within the area of stenosis divided by peak systolic velocity in a normal adjacent proximal artery segment) in the treated segment at 12 months after intervention as determined by catheter angiography or Duplex ultrasound.

SECONDARY OUTCOMES:
Limb salvage rate free of above-the-ankle amputation. | One year
Sustained clinical improvement rate. | One year
Repeated target lesion revascularization (TLR) rate. | One year
Repeated target extremity revascularization (TER) rate. | One year
Total reocclusion rate. | One year
Comparison of late angiographic restenosis (%). | One year
Ankle-brachial index (ABI). | One year
The rate of major adverse cardiovascular events (MACE) composed of all-cause death, myocardial infarction and stroke. | One year
The duration of the procedure from just before the guidewire enters the lesion, to when it proceeds into the distal normal vessel | One year
The amount of contrast from just before the guidewire enters the lesion, to when it proceeds into the distal normal vessel | One year
The length of distal normal vessel's injury related to the guidewire or re-entry device. | One year
Incidence of vascular perforation with the failure rate of procedure. | One year
Death rate related to procedure. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Woon Rha, MD, PhD, Principal Investigator — Cardiovascular Center, Korea University Guro Hospital, 80, Guro-dong, Guro-gu, Seoul, 152-703, South Korea
Locations (3):
- South Korea (3):
  - Cardiovascular center, Korea University Guro Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seung Woon Rha, Seoul

REFERENCES:
- [Background] Bolia A, Miles KA, Brennan J, Bell PR. Percutaneous transluminal angioplasty of occlusions of the femoral and popliteal arteries by subintimal dissection. Cardiovasc Intervent Radiol. 1990 Dec;13(6):357-63. doi: 10.1007/BF02578675. PMID 2149672
- [Background] Noory E, Rastan A, Sixt S, Schwarzwalder U, Leppannen O, Schwarz T, Burgelin K, Hauk M, Branzan D, Hauswald K, Beschorner U, Nazary T, Brantner R, Neumann FJ, Zeller T. Arterial puncture closure using a clip device after transpopliteal retrograde approach for recanalization of the superficial femoral artery. J Endovasc Ther. 2008 Jun;15(3):310-4. doi: 10.1583/07-2324.1. PMID 18540697
- [Background] Montero-Baker M, Schmidt A, Braunlich S, Ulrich M, Thieme M, Biamino G, Botsios S, Bausback Y, Scheinert D. Retrograde approach for complex popliteal and tibioperoneal occlusions. J Endovasc Ther. 2008 Oct;15(5):594-604. doi: 10.1583/08-2440.1. PMID 18840044
- [Background] Bosiers M, Deloose K, Callaert J, Maene L, Keirse K, Verbist J, Peeters P. In lower extremity PTAs intraluminal is better than subintimal. J Cardiovasc Surg (Torino). 2012 Apr;53(2):223-7. PMID 22456645
- [Background] Soga Y, Iida O, Suzuki K, Hirano K, Kawasaki D, Shintani Y, Suematsu N, Yamaoka T. Initial and 3-year results after subintimal versus intraluminal approach for long femoropopliteal occlusion treated with a self-expandable nitinol stent. J Vasc Surg. 2013 Dec;58(6):1547-55. doi: 10.1016/j.jvs.2013.05.107. Epub 2013 Aug 1. PMID 23910456
- [Background] Laird JR, Katzen BT, Scheinert D, Lammer J, Carpenter J, Buchbinder M, Dave R, Ansel G, Lansky A, Cristea E, Collins TJ, Goldstein J, Jaff MR; RESILIENT Investigators. Nitinol stent implantation versus balloon angioplasty for lesions in the superficial femoral artery and proximal popliteal artery: twelve-month results from the RESILIENT randomized trial. Circ Cardiovasc Interv. 2010 Jun 1;3(3):267-76. doi: 10.1161/CIRCINTERVENTIONS.109.903468. Epub 2010 May 18. PMID 20484101
- [Background] Strecker EP, Boos IB, Gottmann D, Vetter S, Haase W. Popliteal artery stenting using flexible tantalum stents. Cardiovasc Intervent Radiol. 2001 May-Jun;24(3):168-75. doi: 10.1007/s002700002526. PMID 11443404
- [Background] Chang IS, Chee HK, Park SW, Yun IJ, Hwang JJ, Lee SA, Kim JS, Chang SH, Jung HG. The primary patency and fracture rates of self-expandable nitinol stents placed in the popliteal arteries, especially in the P2 and P3 segments, in Korean patients. Korean J Radiol. 2011 Mar-Apr;12(2):203-9. doi: 10.3348/kjr.2011.12.2.203. Epub 2011 Mar 3. PMID 21430937
- [Background] Kidd J, Bourke BM, Dunwoodie J et al. The role of pre and postprocedural color Duplex ultrasound for the treatment of lower limb ischemia by subintimal angioplasty. J Vasc Ultrasound. 2006;30:17-21.
- [Background] Lipsitz EC, Ohki T, Veith FJ, Suggs WD, Wain RA, Cynamon J, Mehta M, Cayne N, Gargiulo N. Does subintimal angioplasty have a role in the treatment of severe lower extremity ischemia? J Vasc Surg. 2003 Feb;37(2):386-91. doi: 10.1067/mva.2003.20. PMID 12563211
- [Background] London NJ, Srinivasan R, Naylor AR, Hartshorne T, Ratliff DA, Bell PR, Bolia A. Reprinted article "Subintimal angioplasty of femoropopliteal artery occlusions: the long-term results". Eur J Vasc Endovasc Surg. 2011 Sep;42 Suppl 1:S9-15. doi: 10.1016/j.ejvs.2011.06.018. PMID 21855032
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Background] Diehm N, Baumgartner I, Jaff M, Do DD, Minar E, Schmidli J, Diehm C, Biamino G, Vermassen F, Scheinert D, van Sambeek MR, Schillinger M. A call for uniform reporting standards in studies assessing endovascular treatment for chronic ischaemia of lower limb arteries. Eur Heart J. 2007 Apr;28(7):798-805. doi: 10.1093/eurheartj/ehl545. Epub 2007 Feb 22. PMID 17317699
- [Background] Duda SH, Pusich B, Richter G, Landwehr P, Oliva VL, Tielbeek A, Wiesinger B, Hak JB, Tielemans H, Ziemer G, Cristea E, Lansky A, Beregi JP. Sirolimus-eluting stents for the treatment of obstructive superficial femoral artery disease: six-month results. Circulation. 2002 Sep 17;106(12):1505-9. doi: 10.1161/01.cir.0000029746.10018.36. PMID 12234956
- [Background] Vollmar J (1975) Rekonstruktive Chirurgie der Arterien. Georg Thieme Verlag, Stuttgart, pp 265-266.